CLINICAL TRIAL: NCT01972373
Title: Visualization of a VEGF-targeted Optical Fluorescent Imaging Tracer in Rectal Cancer During Flexible NIR Fluorescence Endoscopy
Brief Title: Visualization of Rectal Cancer During Endoscopy, Using a Fluorescent Tracer
Acronym: RAPIDO-TRACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL43407.042.13; 2013-000333-12 (EudraCT Number)
Record Dates: First submitted 2013-10-21; First posted 2013-10-30 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer
Keywords: VEGF; Fluorescence; Endoscopy; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NIR endoscopy with Bevacizumab-IRDye800CW (Experimental): In this non-randomized, non-blinded, prospective, feasibility study, bevacizumab-IRDye800CW will be administered to a total of 30 patients with proven locally advanced rectal cancer.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: NIR fluorescence endoscopy

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — Intravenous administration of a microdose (4.5mg, subtherapeutic) of Bevacizumab-IRDye800CW prior to the endoscopic procedure
  Other Names: Fluorescence tracer imaging; Beva-800CW; Bevacizumab-800CW
Device: NIR fluorescence endoscopy — 48-72 hours administration of Bevacizumab-IRDye800CW a flexible NIR fluorescence endoscopy will be performed via the rectum
  Other Names: Sigmoid endoscopy using near infrared fluorescence

SUMMARY:
To improve rectal cancer management, there is a need for better visualization of drug targets in rectal cancer to identify patients who might benefit from specific targeted treatments. Molecular imaging of rectal cancer associated targets is a promising technique to accommodate this need. Vascular Endothelial Growth Factor (VEGF), which is differentially expressed in normal versus malignant colon tissue, has proven to be a valid target for molecular imaging. Fluorescent labeling of bevacizumab (a VEGF targeting humanized monoclonal antibody currently used in anti-cancer therapy) using IRDye800CW (a fluorescent dye) has potential advantages in view of safety, infrastructure, costs, stability and imaging resolution. Therefore, the fluorescent tracer bevacizumab-IRDye800CW has been developed at the University Medical Center Groningen (UMCG) and was recently approved to be administered to patients in a tracer dose. To detect this tracer in vivo in patients with colorectal cancer, a newly developed flexible near-infrared (NIR) fluorescence endoscope and optoacoustic endoscope have been developed which can be used in clinical studies. Optical fluorescence imaging may support response evaluation following chemoradiotherapy and give insight which patient might benefit from anti-VEGF targeted therapy in future studies.

DETAILED DESCRIPTION:
In this non-randomized, non-blinded, prospective, single center feasibility study, patients with locally advanced rectal cancer who are included in the RAPIDO study (NL36315.042.11) will undergo two times epi-illumination endoscopy (in other words flexible NIR fluorescence endoscopy).

The study consists of a total of five study procedure related visits:

* Visit 1: During a screening visit, eligibility will be evaluated and patient characteristics will be collected.
* Visit 2: During the second visit 4.5 mg of bevacizumab-IRDye800CW will be administered intravenously. The patient will then be observed for 1 hour post administration.
* Visit 3: First endoscopy will be performed at baseline (two days after tracer administration); before the start of chemoradiotherapy.
* Visit 4: After chemoradiotherapy patients will receive a second dose of 4.5 mg of bevacizumab-IRDye800CW (second tracer administration)
* Visit 5: A second flexible NIR fluorescence endoscopy procedure will be performed (two-three days after the second tracer injection), preferably right before surgery.

Optionally and when available, we will ask patients if they would like to undergo optoacoustic endoscopy. This is a form of endoscopic ultrasound which is able to detect bevacizumab-IRDye800CW up to 2 cm in depth. The procedure is comparable with NIR fluorescence endoscopy. If patients agree, after removal of the NIR fluorescence endoscope the optoacoustic endoscope will be introduced in the rectum of the patient for detection of bevacizumab-IRDye800CW in deeper areas of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven, newly diagnosed primary rectal adenocarcinoma, i.e. with the lowest part of the tumor less than 16 cm from the anal verge using a rigid rectoscope or flexible endoscope.
* Locally advanced tumor fulfilling at least one of the following criteria on pelvic MRI indicating high risk of failing locally and/or systemically:

  * Clinical stage (c)T4a
  * cT4b
  * Extramural vascular invasion (EMVI+)
  * N2 i.e. four or more lymph nodes in the mesorectum showing morphological signs on MRI indicating metastatic disease
  * positive mesorectal fascia (MRF), i.e. tumor or lymph node one mm or less from the mesorectal fascia
  * metastatic lateral nodes, > 1 cm (lat Lymph Node+)
* Staging done within 5 weeks before randomization.
* No contraindications to chemotherapy, including adequate blood counts:

  * White blood count ≥4.0 x 109/L;
  * Platelet count ≥100 x 109/L;
  * Clinically acceptable haemoglobin levels;
  * Creatinine levels indicating renal clearance of ≥50 ml/min;
  * Bilirubin <35 μmol/l
* Eastern Cooperative Oncology Group (ECOG) performance score < 1.
* Patient is considered to be mentally and physically fit for chemotherapy as judged by the medical oncologist.
* Age ≥ 18 years.
* Written informed consent.
* Adequate potential for follow-up.

Exclusion Criteria:

* Extensive growth into cranial part of the sacrum (above S3) or the lumbosacral nerve roots indicating that surgery will never be possible even if substantial tumour down-sizing is seen.
* Presence of metastatic disease or recurrent rectal tumour. Familial Adenomatosis Polyposis coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active ulcerative Colitis.
* Concomitant malignancies, except for adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri. Subjects with prior malignancies must be disease-free for at least 5 years.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Any contraindications to MRI (e.g. patients with pacemakers).
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Concurrent uncontrolled medical conditions.
* Any investigational treatment for rectal cancer within the past month.
* Pregnancy or breast feeding.
* Patients with known malabsorption syndromes or a lack of physical integrity of the upper gastrointestinal tract.
* Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac dysrhythmia, e.g. atrial fibrillation, even if controlled with medication) or myocardial infarction within the past 12 months.
* Patients with symptoms or history of peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the marker bevacizumab-IRDye800CW | First endoscopic procedure before start radio-chemotherapy and second endoscopic procedure 3 weeks after start of radiochemotherapy
  To determine the sensitivity of the marker bevacizumab-IRDye800CW measured by innovative molecular imaging flexible NIR fluorescence endoscopy, and optionally optoacoustic endoscopy, in identifying target expression and heterogeneity prior to the start, or during early treatment, of neoadjuvant radiochemotherapy, to identify patients who benefit from additional treatment targeting VEGF to increase pCR in future studies.
  Research aim to assess primary objectives by evaluation of biopsy specimen:
  * To assess accumulation of bevacizumab-IRDye800CW in rectal cancer tissue and surrounding tissue at baseline and following radiochemotherapy of patients included in the RAPIDO trial.
  * Evaluation of tumor areas with high fluorescence and low fluorescence signal.
  * To correlate the above to VEGF-levels determined by immuno-histochemistry.

SECONDARY OUTCOMES:
Correlation between bevacizumab-IRDye800CW uptake and pathological response (pCR) | Endoscopic procedures before and after chemoradiation therapy, assesing of pathological respons after churgical intervention
In vivo quantification of the NIR fluorescent signal of bevacizumab-IRDye800CW using the NIR fluorescence endoscope vs. ex vivo VEGF levels in biopsies | Before start and after chemoradiation therapy
To Perform correlate pathways analyses using RNA/DNA/protein analyses to NIR fluorescence data | After surgery
The ability of optoacoustic endoscopy to detect bevacizumab-IRDye800CW in deeper areas of the tumor | Before start and after chemoradiation therapy
Collection of safety regarding administration of Bevacizumab-IRDye800CW | Participants will be followed the duration of the chemoradiation therapy till surgery
  To abtain information on safety aspectsof the tracer, side effects, adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR)

CONTACTS AND LOCATIONS:
Overall Officials: Wouter B Nagengast, MD, PhD, Principal Investigator — University Medical Center Groningen; Geke AP Hospers, Prof. dr., Principal Investigator — University Medical Center Groningen; Boudewijn v. Etten, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] de Jongh SJ, Tjalma JJJ, Koller M, Linssen MD, Vonk J, Dobosz M, Jorritsma-Smit A, Kleibeuker JH, Hospers GAP, Havenga K, Hemmer PHJ, Karrenbeld A, van Dam GM, van Etten B, Nagengast WB. Back-Table Fluorescence-Guided Imaging for Circumferential Resection Margin Evaluation Using Bevacizumab-800CW in Patients with Locally Advanced Rectal Cancer. J Nucl Med. 2020 May;61(5):655-661. doi: 10.2967/jnumed.119.232355. Epub 2019 Oct 18. PMID 31628218
- [Derived] Tjalma JJJ, Koller M, Linssen MD, Hartmans E, de Jongh SJ, Jorritsma-Smit A, Karrenbeld A, de Vries EG, Kleibeuker JH, Pennings JP, Havenga K, Hemmer PH, Hospers GA, van Etten B, Ntziachristos V, van Dam GM, Robinson DJ, Nagengast WB. Quantitative fluorescence endoscopy: an innovative endoscopy approach to evaluate neoadjuvant treatment response in locally advanced rectal cancer. Gut. 2020 Mar;69(3):406-410. doi: 10.1136/gutjnl-2019-319755. Epub 2019 Sep 18. No abstract available. PMID 31533965